CLINICAL TRIAL: NCT05648188
Title: Assessing the Expression of A2R Receptors and CD39 and CD73 Ectonucleotidases on Circulating Tumour Cells of Non-small Cell Lung Carcinoma
Brief Title: A2R and Ectonucleotidases Expression in Lung Cancer Circulating Tumor Cells
Acronym: LUNGadenosine
Status: Withdrawn | Type: Observational
Why Stopped: no patients enrolled
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Pneumo01
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (20 ml). tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NSCLC patients: Patients with proven stage IA-IIB non-small cell lung cancer (NSCLC).
  Interventions: Biological: Sample

INTERVENTIONS:
Biological: Sample — Sample of whole blood and tissue for ex vivo expression of A2R, CD39, CD73 and P2RX7

SUMMARY:
Early non-small cell lung cancer (NSCLC), treated by surgery or radiotherapy in the case of inoperability, relapses in almost 50% of cases. Circulating tumour cells (CTCs), which can be detected before surgery, represent a promising prognostic tool, but the markers characterising their aggressiveness remain to be determined. The NSCLC microenvironment, in which purinergic signalling is a key pathway, controls tumour development. Adenosine derived from the action of CD39 and CD73 ectonucleotidases hydrolysing extracellular ATP, induces immunosuppression of NSCLC by activating A2R receptors. The expression and prognostic relevance of A2R, CD39 and CD73 on CTCs is unknown. The objectives are to (i) compare the expression of A2R and CD39 and CD73 on primary tumour cells and CTCs of patients operated on for early NSCLC, (ii) correlate these data with molecular characteristics and clinical response, (iii) determine on lung cancer lines whether irradiation impacts on the expression of A2R, CD39 and CD73. This work could contribute to the identification of new theranostic biomarkers.

ELIGIBILITY:
i) Inclusion criteria:

* Patient of legal age (>18 years), any gender,
* operated on for stage (IA to IIB) non-small cell lung cancer (NSCLC)

ii) Exclusion criteria:

* Patient with any other active cancer.
* Lack of evaluable material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for a localized NSCLC (IA-IIB stage) in Nice University Hospital, Thoracic Surgery service.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Ex vivo expression of A2R (adenosine receptor), CD39, CD73 and P2RX7 on NSCLC and CTC | At inclusion
  Presence versus Absence of expression (immunohistochemistry)

SECONDARY OUTCOMES:
In vitro impact of radiation therapy on the A2R, CD39, CD73 expression by cells lineage | At inclusion
  Upregulation / Downregulation of expression (mRNA by real time PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan BENZAQUEN, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No